CLINICAL TRIAL: NCT07163338
Title: A Prospective, Single-center Cohort Study to Determine the Prevalence and Consequences of Antiphospholipid Syndrome in Patients Aged 65 and Over With Ischemic Strokes (IS)
Brief Title: Prevalence and Consequences of Antiphospholipid Syndrome in Patients Aged 65 and Over With Ischemic Strokes (IS)
Acronym: SAPLAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PL25066
Record Dates: First submitted 2025-06-27; First posted 2025-09-09 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-06

CONDITIONS: Antiphospholipid Syndrome
Keywords: Antiphospholipid syndrome; antiphospholipid antibody syndrome; stroke; ischemic stroke
MeSH Terms: conditions — Antiphospholipid Syndrome; Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Other: Collectio nof blood

INTERVENTIONS:
Other: Collectio nof blood — Collection of an additional volume of blood in the initial blood test.

SUMMARY:
Stroke represents a major cause of morbidity and mortality despite significant progress in recent decades. In individuals under the age of 65, the etiologies of ischemic stroke (IS) are diverse, and management is well-established. Antiphospholipid syndrome (APS) accounts for 10 to 20% of the causes of stroke in this population. In elderly individuals, APS is not systematically investigated due to the predominance of embolic, atherosclerotic, and small vessel disease causes. However, delayed discovery of APS is not uncommon and is more frequently associated with the occurrence of arterial thrombosis. Moreover, the management of APS involves several challenges given the risk of recurrence of thrombosis and the potential association with conventional cardiovascular risk factors. The antithrombotic treatment consists of lifelong anticoagulation, excluding direct oral anticoagulants (DOACs) due to the risk of thrombotic recurrence. The main objective of the study will be to assess the prevalence of antibodies useful for the diagnosis of APS (Sapporo criteria) in individuals aged 65 or older hospitalized for an ischemic stroke (IS) or transient ischemic attack (TIA).

Furthermore, the classification of APS is likely to evolve in the coming years with the inclusion of new clinically relevant antibodies (anti-phosphatidylserine and anti-phosphatidylethanolamine) because of their strong association with the occurrence of thrombosis. Even though they are often associated with circulating anticoagulants, they are also found in 10% of APS cases negative for other antibodies.

Patient inclusion in the study should occur during the acute phase of the stroke, before the initiation of anticoagulant treatment.

Thus, after verifying the inclusion and exclusion criteria, patients will be informed and must sign the informed consent form if they agree to participate.

After inclusion, the research procedure will be as follows:

* Conduct a unique immunological biological assessment with:

  * Part performed as part of standard care: circulating anticoagulants, anti-cardiolipin antibodies, and anti-β2-glycoprotein type 1.
  * Part performed specifically for the study (3.5 mL of additional blood): anti-phosphatidylserine and anti-phosphatidylethanolamine antibodies. The search for these antibodies will be performed using the 7mL dry tube collected for anti-cardiolipin and anti-β2-glycoprotein type 1 antibody testing.
  * If the diagnostic sample is positive for any of these antibodies, a follow-up at 3 months is recommended and will be performed as part of standard care to confirm the APS diagnosis.
* Data collection will include patient details, stroke/TIA details, biological data, and follow-up. As part of routine follow-up, patients will be seen in a neurological consultation at 6 months.

Clinical and biological data will be reviewed at the end of the study by two doctors (a neurologist and an internist) to confirm or exclude the APS diagnosis and its contribution to the neurological condition.

An internal medicine follow-up will be initiated for patients with confirmed APS, and an appropriate treatment will be proposed.

DETAILED DESCRIPTION:
Stroke represents a major cause of morbidity and mortality despite significant progress in recent decades, particularly in acute-phase management. In 80% of cases, stroke is ischemic (IS), and the etiology and prognosis can vary depending on the patient's age. A comprehensive etiological workup allows for the adaptation of secondary prevention, thereby helping to reduce the risk of recurrence.

In individuals under the age of 65, etiologies of ischemic stroke (IS) are multiple, and management is well-established. In individuals under 50, antiphospholipid syndrome (APS) accounts for 10 to 20% of the causes of ischemic stroke, highlighting the importance of this etiology in younger patients. The diagnosis of IS/TIA related to APS relies on expert evaluation of clinical and biological data.

This syndrome is characterized by thrombosis in arterial or venous territories as well as the detection of specific antibodies (anti-cardiolipin antibodies, and/or anti-β2-glycoprotein type 1 antibodies, and/or circulating anticoagulants), with a cumulative risk of thrombosis depending on the number of antibodies identified. Historically, APS was associated with lupus and considered secondary, but it is now well accepted that it can occur in isolation and thus be primary.

APS is not systematically sought in elderly patients due to the predominance of cardioembolic, atherosclerotic, and small vessel disease causes. However, the late discovery of APS is not uncommon and is more frequently associated with arterial thrombosis. A retrospective study including a systematic search for APS in patients with IS found a significant association between older age and the presence of antiphospholipid antibodies (71 vs 66 years). Management presents several challenges due to the risk of recurrence of both arterial and venous thrombosis, as well as the potential association with conventional cardiovascular risk factors. Antithrombotic treatment involves lifelong anticoagulation, excluding direct oral anticoagulants (DOACs) such as Rivaroxaban due to the risk of thrombotic recurrence. A retrospective study also showed an association between APS and atrial fibrillation, reaching 30%. Atrial fibrillation, the prevalence of which increases with age, is increasingly treated with DOACs, suggesting the need to investigate APS in order to adapt the antithrombotic treatment and reduce the risk of recurrence.

Furthermore, the classification of APS is likely to evolve in the coming years with the inclusion of new clinically relevant antibodies, such as anti-phosphatidylserine and anti-phosphatidylethanolamine. These antibodies are strongly associated with the occurrence of thrombosis. Moreover, although these antibodies are strongly associated with circulating anticoagulants (which are difficult to detect due to the need for no anticoagulant treatment at the time of sample collection), they are also found in 10% of APS cases that are negative for other antibodies. With this study, we propose to systematically investigate these two antibodies as well.

Patient inclusion in the study should occur during the acute phase of the stroke, before the initiation of anticoagulant treatment.

Thus, after verifying the inclusion and exclusion criteria:

* If the patient's condition allows, the patient will be informed of the study's methods and objectives and must sign the informed consent form if they agree to participate.
* If the patient's condition does not permit informing them or obtaining their consent, close relatives present will be informed about the study's objectives and methods and will be asked to sign the consent form if they agree to the patient's participation. The patient will be informed as soon as possible, and their consent will be requested for continued participation if needed.

After inclusion, the research procedure will be as follows:

* Conduct a unique immunological biological assessment with:

  * Part performed as part of standard care: circulating anticoagulants, anti-cardiolipin antibodies, and anti-β2-glycoprotein type 1.
  * Part performed specifically for the study (3.5 mL of additional blood): anti-phosphatidylserine and anti-phosphatidylethanolamine antibodies. The search for these antibodies will be performed using the 7mL dry tube collected for anti-cardiolipin and anti-β2-glycoprotein type 1 antibody testing.
  * If the diagnostic sample is positive for any of these antibodies, a follow-up at 3 months is recommended and will be performed as part of standard care to confirm the APS diagnosis.
* Data collection will include patient details (age, sex, etc.), stroke/TIA (location, etiology, etc.), biological data, and follow-up (recurrence, disability, and mortality during hospitalization and at 6 months). As part of routine follow-up, patients will be seen in a neurological consultation at 6 months.

Clinical and biological data will be reviewed at the end of the study by two doctors (a neurologist and an internist) to confirm or exclude the APS diagnosis and its contribution to the neurological condition.

An internal medicine follow-up will be initiated for patients with confirmed APS, and an appropriate treatment will be proposed.

ELIGIBILITY:
inclusion criteria :

* patients aged 65 and over during the inclusion phase
* hospitalized for a TIA/ischemic stroke in neurology or internal medicine department during the inclusion phase
* affiliated with social security system exclusion criteria :
* patients under 65 years old
* under legal guardianship, curatorship, or tutorship
* incarcerated
* under psychiatric care
* admitted to a healthcare or social institution

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-12-16 (Estimated); Study Completion 2028-03-16 (Estimated)

PRIMARY OUTCOMES:
Prevalence of antiphospholipid antibodies in patients aged at least 65 years hospitalized for a TIA or an ischemic stroke | At the inclusion
  Evaluate the prevalence of antibodies useful for the diagnosis of Antiphospholipid syndrome in patients aged at least 65 years hospitalized for a TIA or a stroke : anticardiolipin antibodies, anti-beta-2-glycoprotein-I lantibodies and lupus anticoagulant

SECONDARY OUTCOMES:
Prevalence of confirmed Antiphospholipid syndrome at 12 weeks | At 12 weeks
  Prevalence of confirmed Antiphospholipid syndrome according to Sapporo criteria
Type of TIA/stroke, location and clinical manifestations | At the inclusion
  In cases of confirmed Antiphospholipid syndrome, describe the type of stroke/TIA, its location and its clinical manifestations
Prevalence of anti-phosphatidylethanolamine antibodies | At the inclusion
  Prevalence of anti-phosphatidylethanolamine antibodies
Prevalence of anti-phosphatidylserine antibodies | At the inclusion
  Prevalence of anti-phosphatidylserine antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France